CLINICAL TRIAL: NCT00675610
Title: Enhancing Communication and HIV Outcomes
Acronym: ECHO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mary Catherine Beach, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ECHO-01; 290-01-0012
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: communication; HIV/AIDS; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Communication; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual care (No Intervention): providers are not trained and patients are not coached
- intervention arm (Experimental): providers are trained to communicate with patients about adherence and patients are coached to discuss adherence with providers
  Interventions: Behavioral: communication training

INTERVENTIONS:
Behavioral: communication training — providers are trained to communicate with patients about adherence and patients are coached to discuss adherence with providers
  Arms: intervention arm

SUMMARY:
The goal of this research is to improve communication between the patients with HIV and their health care providers. The overall purpose of doing so is to reduce disparities in medication self-efficacy, adherence to therapy, and HIV viral load suppression. The investigators will conduct a randomized controlled trial to test the effectiveness of a combined provider and patient communication intervention conducted at two separate visits compared to usual care in improving the quality of patient-provider communication, patients' medication self-efficacy, patient adherence to therapy, and HIV RNA suppression.

DETAILED DESCRIPTION:
The goal of this research is to improve communication between the patients with HIV and their health care providers. The overall purpose of doing so is to reduce disparities in medication self-efficacy, adherence to therapy, and HIV viral load suppression. We will conduct a randomized controlled trial to test the effectiveness of a combined provider and patient communication intervention conducted at two separate visits compared to usual care in improving the quality of patient-provider communication, patients' medication self-efficacy, patient adherence to therapy, and HIV RNA suppression. The following primary and secondary hypotheses will be addressed.

Primary Hypothesis.

1) There will be more and higher quality patient-provider communication about antiretroviral medication adherence in the intervention compared to control arm at both visit 1 (V1) and visit 2 (V2).

Secondary Hypotheses

1. Higher quality patient-provider communication in the intervention arm will be associated with

   * higher patient ratings of communication (overall, HIV-specific, adherence-specific, and interpersonal style of provider) at V1 and V2;
   * increased patient preference for a shared decision-making role at V1 and V2;
   * more positive health beliefs at V1 and V2;
   * higher patient medication self-efficacy at V1 and V2;
   * better adherence to antiretroviral medication (assessed by 3-day recall) at V2; and
   * a greater percentage of patients with HIV-1 RNA suppression at V2.
2. The intervention will reduce disparities in medication self-efficacy, adherence, and HIV-1 RNA suppression.

ELIGIBILITY:
Inclusion Criteria (Providers):

1. Currently providing primary care to at least 10 HIV-infected patients in the clinic
2. Physician, Nurse-Practitioner, or Physician-Assistant
3. Agree to give written informed consent.

Inclusion Criteria (Patients):

1. HIV-infected patient of one of the participating providers
2. Has had at least one prior visit with that provider
3. Currently taking antiretroviral therapy
4. Capable of understanding and giving written informed consent
5. Age > 20 years old
6. English-speaking
7. African-American (or people of African descent living in the United States), Hispanic, or non-Hispanic White race/ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
patient-provider communication | 1 day- 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Catherine Beach, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - Wayne State University, Detroit, Michigan
  - Saint Lukes-Roosevelt, New York, New York
  - Oregon Health Science University, Portland, Oregon